CLINICAL TRIAL: NCT07231601
Title: Laparoscopic Mesenteric Excision and Exclusion for Crohn's Disease of the Terminal Ileum. A Greek Single Center Study.
Brief Title: Laparoscopic Right Hemicolectomy for Crohn's Disease of the Terminal Ileum Utilizing the Mesenteric Excision and Exclusion
Status: Recruiting | Type: Observational
Sponsor: Tzaneio General Hospital (Other)
Responsible Party: Principal Investigator, Panagiotis Dikeakos, Consultant, Tzaneio General Hospital
Other Study IDs: 15094- 23/09/2025
Record Dates: First submitted 2025-08-31; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Crohn Disease (CD); Crohn Disease of Ileum; Kono S Anastomosis; Extended Mesenteric Excision
Keywords: Kono-s; extended mesenteric excision; mesenteric excision and exclusion
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Crohn's disease of the terminal ileum: Patients with Crohn's disease of the terminal ileum requiring surgical intervention
  Interventions: Procedure: Mesenteric excision and exclusion

INTERVENTIONS:
Procedure: Mesenteric excision and exclusion — Laparoscopic segmental right colectomy and excision of the affected terminal ileum with extended mesenteric excision and open Kono-s anastomosis

SUMMARY:
This study is designed for patients requiring surgery for Crohn's disease of the terminal ileum. A combination of laparoscopic segmental right colectomy with extended mesenteric excision and the Kono-s anastomosis will be utilized. Since this is a fairly new technique, the intra and post operative complications will be reviewed. Also endoscopic, clinical and surgical reoccurrence will be reviewed at certain predefined time points post operatively.

DETAILED DESCRIPTION:
Crohn's disease is a chronic inflammatory disease that can affect any part of the gastrointestinal tract. The underlying etiology is still unknown, but it is perceived multifactorial and the effect of environmental and pathophysiological factors on a genetically predisposed individual.

Although the development of new pharmacological agents has revolutionized the management of Crohn's disease, the rates of endoscopic and surgical reoccurrence still remain discouraging. It is estimated that 50% of patients with Crohn's disease will require surgical intervention and the rate of surgical reoccurrence remains as high as 30% at 10 years.

Since most reoccurrences occur near or around the anastomotic site, the type of resection and anastomosis has been extensively reviewed in the past, but no significant differences have been observed. In the later years two new surgical techniques have been developed (extended mesenteric excision and Kono-S anastomosis), and increasing data show that they could potentially reduce the rate of reoccurrence. Both techniques focus on the role of the mesentery on disease reoccurrence. The extended mesenteric excision removes the mesentery and corresponding lymphatics of the affected bowel while the Kono-S anastomosis excludes the mesentery from the overlying wide anastomosis. The combination of the two techniques has been termed "mesenteric excision and exclusion" The primary goal of this study is to assess the safety the mesenteric excision and exclusion for Crohn's diseases disease of the terminal ileum in a central hospital of Greece. All intra and postoperative complications within 30 days will be collected and reviewed.

As secondary goals, the endoscopic, clinical and surgical reoccurrence will be reviewed at 6 months, 2 years and 5 years after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged >16 years
* Ileocolic disease or disease of the terminal ileum with an indication for resection
* Concurrent therapies with corticosteroids, 5-ASA drugs, thiopurines, MTX, antibiotics, and anti-TNF therapy are permitted.
* All patients should have undergone a colonoscopy and a recent update of imaging (e.g. Ultrasound, MR enterography (or CT enterography if MR is contraindicated))
* Ability to comply with protocol.
* Competent and able to provide written informed consent.

Exclusion Criteria:

* Inability to give informed consent.
* Patients less than 16 years of age.
* Clinically significant medical conditions within the six months before the operation : e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the patient.
* History of cancer < 5 years which might influence patients prognosis
* Emergent operation.
* Pregnant or breast feeding.
* Inability to follow up at 3, 6 and 12 months for postoperative assessment, imaging and endoscopy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Community based study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of the procedure | 30 days post intervention
  Collection of intra and post operative complication rate

SECONDARY OUTCOMES:
Endoscopic reoccurence | 6 months, 2 years and 5 years post intervention
  Endoscopic reoccurrence according to Rutgeert's score
Clinical reoccurrence | Up to 5 years
  Clinical symptoms severe enough to require new endoscopy
Surgical reoccurrence | Up to 5 years
  Repeat surgery because of reoccurrence at the proximity of the Kono-S anastomosis

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Ayiomamitis, Study Director — General Hospital of Piraeus "Tzaneio"
Locations (1):
- General Hospital Of Piraeus "Tzaneio", Piraeus, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Patient Characteristics
Supporting Information: ICF
Time Frame: 01/01/2022- 31/12/2032
Access Criteria: The information is freely available
URL: https://figshare.com/articles/dataset/Mesenteric_excision_and_exclusion_for_ileocolic_Crohn_s_disease_A_Greek_single_center_study_/30084286?file=57789025

REFERENCES:
- [Background] Kono T, Fichera A, Maeda K, Sakai Y, Ohge H, Krane M, Katsuno H, Fujiya M. Kono-S Anastomosis for Surgical Prophylaxis of Anastomotic Recurrence in Crohn's Disease: an International Multicenter Study. J Gastrointest Surg. 2016 Apr;20(4):783-90. doi: 10.1007/s11605-015-3061-3. Epub 2015 Dec 22. PMID 26696531
- [Background] Coffey CJ, Kiernan MG, Sahebally SM, Jarrar A, Burke JP, Kiely PA, Shen B, Waldron D, Peirce C, Moloney M, Skelly M, Tibbitts P, Hidayat H, Faul PN, Healy V, O'Leary PD, Walsh LG, Dockery P, O'Connell RP, Martin ST, Shanahan F, Fiocchi C, Dunne CP. Inclusion of the Mesentery in Ileocolic Resection for Crohn's Disease is Associated With Reduced Surgical Recurrence. J Crohns Colitis. 2018 Nov 9;12(10):1139-1150. doi: 10.1093/ecco-jcc/jjx187. PMID 29309546
- [Background] Holubar SD, Gunter RL, Click BH, Achkar JP, Lightner AL, Lipman JM, Hull TL, Regueiro M, Rieder F, Steele SR. Mesenteric Excision and Exclusion for Ileocolic Crohn's Disease: Feasibility and Safety of an Innovative, Combined Surgical Approach With Extended Mesenteric Excision and Kono-S Anastomosis. Dis Colon Rectum. 2022 Jan 1;65(1):e5-e13. doi: 10.1097/DCR.0000000000002287. PMID 34882636